CLINICAL TRIAL: NCT00448084
Title: BOLD-fMRI of the Perception of Volition in Functional Movement Disorders
Brief Title: Brain Activity in People With Functional Movement Disorders
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 070117; 07-N-0117
Record Dates: First submitted 2007-03-14; First posted 2007-03-15 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-08-05

CONDITIONS: Functional Movement Disorders
Keywords: Psychogenic Movement Disorders; Volition; fMRI; Functional MRI; Functional Movement Disorder; Healthy Volunteer; HV
MeSH Terms: conditions — Conversion Disorder; Self-Control

SUMMARY:
This study will use functional MRI (fMRI, a technique that shows what areas of the brain are active when performing different mental tasks), to examine how the brain in people with functional movement disorders (FMD) may differ from that in people without FMDs. People with FMD have movement symptoms they feel they cannot control and that are not due to a known medical disorder. Previous studies looking at the brain activity of FMD patients have found areas in the frontal lobe of the brain that appeared overactive. These overactive areas may make it difficult to perform complex mental tasks. Studying the brain during performance of these tasks may enhance knowledge about FMD.

Patients 18 years of age or older with an FMD and healthy normal volunteers may be eligible for this study. Participants have two visits to the NIH Clinical Center for the following procedures:

First visit (screening):

* Medical history and neurological examination.
* Urine drug screen for illicit drugs.
* Psychological testing, including an interview and questionnaires.

Second visit:

* Brain MRI (if one has not been done at NIH within the past 12 months): MRI uses a magnetic field and radio waves to produce images of body tissues and organs. The subject lies on a table that can slide in and out of the scanner (a narrow cylinder), wearing earplugs to muffle loud noises that occur during the scanning process. The procedure lasts about 2 hours, during which time the patient is asked to lie still for up to 30 minutes at a time.
* Brain fMRI: While in the MRI scanner, subjects read questions and answer them yes or no by pushing buttons. They are asked to answer questions about their health, their movement symptoms and unrelated topics (like personal preferences and current events). The questions vary in difficulty. Sometimes subjects are instructed to answer correctly; other times they are asked to answer incorrectly. A strap is placed around the subject's chest and two wires are taped to the fingers to monitor heart rate, breathing rate and sweat response during the scan. The scan takes about 2 hours.

DETAILED DESCRIPTION:
OBJECTIVE

The purpose of this study is to utilize functional MRI (fMRI) to identify structural brain regions and activation patterns involved in deception in order to determine whether illness deception can be differentiated from involuntary conversion disorders. We intend to compare the brain activations of functional movement disorder (FMD) patients against those of healthy volunteers in order to determine whether various aspects of the disorder are under volitional control, suggesting a component of illness deception, or are involuntary as hypothesized in conversion disorders.

STUDY POPULATION

We intend to use up to 35 right-hand dominant adult healthy volunteers (the first five subjects will be used to develop this method) and 30 functional movement disorder patients.

DESIGN

Using a slow event-related design, we will scan subjects using a 3T fMRI scanner while they are visually presented with survey-based stimuli which require a yes/no response using a key press. Information used to create the stimuli will be pseudo-randomly derived from one of two databases. The first database will be created from the information garnered in the survey subjects will complete during their screening visit (i.e. subjects eye color or height). The second database will be a collection of non-specific information (i.e. current year, season, etc.) that intentionally does not apply to the subjects. For each question displayed, subjects will receive a visual instruction to respond either truthfully or deceptively. Correct answers to responses will be evaluated based upon the survey the subjects completed. In addition to the BOLD data collected, we plan to calculate reaction times and acquire autonomic data in order to identify possible correlates with the brain responses.

OUTCOME MEASURES

The primary outcome measure is the BOLD-fMRI data collected from subjects while answering yes-no type questions. Secondary outcome measures will include reaction times and autonomic data that will be collected simultaneously with the fMRI data. Standard univariate general linear model analysis will be performed on the fMRI data as well as the use of multivariate methods, including support vector machine learning. Subgroup analyses will be conducted to characterize the correlation between reaction times, autonomic data, and fMRI results as well as potential differences in activation patterns for subject-referenced questions and questions which are unrelated to the subject.

ELIGIBILITY:
* INCLUSION CRITERIA:

PATIENTS:

* Age 18 to 65
* Subjects willing to abstain from caffeine or alcohol for 48 hours prior to the fMRI scanning
* Diagnosis of a functional movement disorder confirmed by a study investigator

HEALTHY VOLUNTEERS:

- Age 18 to 65

EXCLUSION CRITERIA:

* Subjects with any abnormal findings on neurological exam consistent with an organic disorder
* Subjects with a positive urine pregnancy test
* Subjects with a positive urine drug screen
* Subjects who are pregnant
* Subjects with any finding on the MRI safety questionnaire which prevents them from safely undergoing an MRI scan
* Subjects with metallic dental fillings which are likely to enhance MRI artifacts
* Subjects with any history of dementia, brain tumor, stroke, head trauma or a vascular malformation as obtained by history or from imaging studies
* Subjects with moderate to severe brain atrophy on imaging studies, as assessed by a study investigator
* Subjects with any history of a severe medical condition, such as cardiovascular disease, which would prevent them from lying flat for up to 120 minutes
* Subjects without the capacity to give informed consent
* Subjects with claustrophobia or other restrictions which prevent them from undergoing a scan in a confined space for up to 120 minutes
* Subjects using beta-blocker medications or other chronotropes which may inhibit the cardiac responsivity
* Patient whose movement frequency and severity prevents them from undergoing MRI safely and effectively for the purposes of data collection
* Patient with a pending medical-legal case
* Subjects with suicidal ideation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65
Dates: Start 2007-03-08; Study Completion 2008-08-05

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Barry RL, Menon RS. Modeling and suppression of respiration-related physiological noise in echo-planar functional magnetic resonance imaging using global and one-dimensional navigator echo correction. Magn Reson Med. 2005 Aug;54(2):411-8. doi: 10.1002/mrm.20591. PMID 16032665
- [Background] Bash IY, Alpert M. The determination of malingering. Ann N Y Acad Sci. 1980;347:86-99. doi: 10.1111/j.1749-6632.1980.tb21257.x. No abstract available. PMID 6930923
- [Background] Cragar DE, Berry DT, Fakhoury TA, Cibula JE, Schmitt FA. Performance of patients with epilepsy or psychogenic non-epileptic seizures on four measures of effort. Clin Neuropsychol. 2006 Sep;20(3):552-66. doi: 10.1080/13854040590947380. PMID 16895866